CLINICAL TRIAL: NCT06553443
Title: Randomised Clinical Trial Comparing Drug-coated Balloon to Plain Balloon for All Peripheral AVF Stenosis
Acronym: RANGER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Singapore Clinical Research Institute (Other); Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RANGER
Record Dates: First submitted 2024-08-11; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Arteriovenous Fistula; Arteriovenous Fistula Stenosis; Dialysis Access Malfunction
Keywords: drug-coated balloon; access circuit patency
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All are blinded except procedurist and protocol administrator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Drug-coated balloon (Experimental): Ranger drug-coated balloon will be used for all peripheral AVF stenosis.
  Interventions: Device: Angioplasty of all peripheral AVF stenosis
- Conventional balloon (Active Comparator): Conventional balloon will be used for all peripheral AVF stenosis.
  Interventions: Device: Angioplasty of all peripheral AVF stenosis

INTERVENTIONS:
Device: Angioplasty of all peripheral AVF stenosis — All peripheral AVF stenosis are to be treated with the same type of balloon depending on allocation

SUMMARY:
To compare the access circuit primary patency after Ranger drug-coated balloon angioplasty of arteriovenous fistula (AVF) stenosis with that after conventional balloon angioplasty

DETAILED DESCRIPTION:
This is a blinded randomized controlled trial recruiting 94 patients with AVF stenosis who will be randomized in a 1:1 ratio to either drug-coated balloon (Ranger) or conventional balloon. All peripheral AVF stenoses will be treated with the allocated balloon type.

The primary outcome measure is 6-month access circuit patency.

ELIGIBILITY:
Inclusion Criteria:

1. Failing AVF with at least 1 AVF stenosis presenting with any clinical, physiological or haemodynamic abnormalities. Both de novo and recurrent stenosis are accepted.
2. AVF has been used successfully for at least 1 month (non-mature AVF are not allowed).
3. Less than 30% residual stenosis after angioplasty.
4. ≥ 21 years old
5. Informed and valid consent given.

Exclusion Criteria:

1. Thrombosed AVFs
2. Haemodynamically significant central vein stenosis
3. Target lesion not treatable with the available sizes of drug eluting balloon (up to 8mm)
4. Contraindication to antiplatelet therapy
5. Coagulopathy or thrombocytopenia that cannot be managed adequately with periprocedural transfusion.
6. Allergy / contraindication to paclitaxel.
7. Acute infection over proposed puncture site.
8. Women who are breastfeeding, pregnant * or planning on becoming pregnant during study.
9. Participant with medical conditions, which in the opinion of the investigator may cause noncompliance with protocol.
10. Currently participating in an investigational drug, biologic or device trial that may have an impact on the dialysis access or previous enrolment in this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Access circuit primary patency | 6 months
  Time to next clinically-driven intervention

SECONDARY OUTCOMES:
Access access circuit patency | 12 months
  Time to next clinically-driven intervention
Access circuit assisted primary patency | 6 and 12 months
  Time to next access thrombosis or surgical intervention.
Access circuit secondary patency | 6 and 12 months
  Time to access abandonment or surgical revision / declotting
Procedural complication | 12 months
  Complication related to procedure
Mortality | 12 months and 5 years
  All cause mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2022-12-28): https://cdn.clinicaltrials.gov/large-docs/43/NCT06553443/Prot_000.pdf